CLINICAL TRIAL: NCT00549653
Title: A Randomized, Single Blind, Repeat Dose, Placebo-controlled, Single-period, Parallel Group Study to Investigate the Safety, Tolerability and Potential Pharmacokinetic Interactions Between GW856553 and Rosuvastatin (10mg), When Co-administered in Healthy Adult Male Subjects
Brief Title: A Study Investigating Blood Concentrations Of Rosuvastatin When Co-administered With GW856553 In Healthy Men
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PM1106502
Record Dates: First submitted 2007-10-24; First posted 2007-10-26 (Estimated); Last update posted 2012-06-04 (Estimated); Status verified 2011-06

CONDITIONS: Atherosclerosis; Cardiovascular Disease
Keywords: GW856553,; drug-drug interactions,; rosuvastatin
MeSH Terms: conditions — Atherosclerosis; Cardiovascular Diseases | interventions — 6-(5-((cyclopropylamino)carbonyl)-3-fluoro-2-methylphenyl)-N-(2,2-dimethylprpyl)-3-pyridinecarboxamide

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: GW856553

SUMMARY:
This study is being conducted to provide initial safety and tolerability data as well as to provide PK data on potential interactions when GW856553 and rosuvastatin are co-administered in healthy male adults

ELIGIBILITY:
Inclusion criteria:

* Healthy adult males, 18-55 years of age, inclusive
* 50Kg >body weight <120Kg
* Body Mass Index (BMI): 19-30
* Must be within 20% of the ideal weight based on height and body frame

Exclusion criteria:

* Any medical history or clinically relevant abnormality identified on the screening medical examination, vital sign measurement, 12-lead ECG recording and/or clinical laboratory examination that is deemed by the principal investigator and/or medical monitor to make the subject ineligible for inclusion because of a safety concern.
* Subjects with rheumatoid arthritis, connective tissue disorders and other conditions known to be associated with chronic inflammation (e.g. Inflammatory Bowel Disease).
* Positive HIV antibody, Hepatitis B surface antigen, Hepatitis C antibody, or other chronic hepatic disorders at screening.
* Subjects with chronic infections such as gingivitis, periodontitis, prostatitis, gastritis, urinary track infections, or any active diseases, including tuberculosis or a history of active tuberculosis.
* Subjects with any acute infection, symptoms suggestive of sinusitis or significant trauma (burns, fractures).
* History of alcohol consumption exceeding, on average, 14 drinks/week for men (1 drink = 5 ounces of wine or 12 ounces of beer or 1.5 ounces of 80 proof distilled spirits) within 6 months of screening.
* Positive urine drug (including cotinine) and/or alcohol at screening.
* A history of smoking within the 3 months prior to screening.
* Use of prescription or non-prescription drugs, including (but not limited to) vitamins, herbal and dietary supplements (including St. John's Wort) within 7 days (or 14 days if the drug is a potential drug inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication. An exception is acetaminophen which is allowed at doses of ≤ 2g/day.
* Participation in a clinical study where the subject has received a drug or new chemical entity within 30 days or 5 half-lives, or twice the duration of the biological effect of any drug (whichever is longer) prior to the first dose of study medication.
* The subject has been exposed to more than four new chemical entities within 12 months prior to the first day of dosing.
* Consumption of any fruit juices (including grapefruit juice) within 7 days prior to the first dose of study medication.
* A history of cholecystectomy or biliary tract disease including a history of liver disease with elevated liver function tests of known or unknown etiology.
* History of increased liver function tests (ALT, AST) above upper limit of normal in the past 6 months and/or liver function tests (bilirubin, ALT, AST) above upper limit of normal at Screening.
* A known history of Gilbert's Syndrome.
* History of myopathy or rhabdomyolysis.
* QTc interval > 450msec.
* An unwillingness of male subjects to abstain from sexual intercourse with pregnant or lactating women; or an unwillingness of the male subject to use a condom/spermicide in addition to having their female partner use another form of contraception, such as: an intrauterine devise (IUD), diaphragm with spermicide, oral contraceptives, injectable progesterone, subdermal implants or a tubal ligation, if the woman could become pregnant from the first dose of study medication until completion of follow-up procedures.
* Donation of blood in excess of 500 mL within 56 days prior to dosing.
* History of sensitivity to heparin or heparin-induced thrombocytopenia.
* Hypersensitivity to rosuvastatin or any component of the rosuvastatin formulation utilised in this study.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2007-10; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
PK blood draws at days 14 and 28 | days 14 and 28

SECONDARY OUTCOMES:
The primary pharmacokinetic endpoints of interest are AUC(0-τ) and Cmax for rosuvastatin | days 14, 15, 28
The secondary pharmacokinetic endpoints of interest are Tmax and t1/2 for rosuvastatin | days 14, 15, 28
Measurement of alanine aminotransferase (ALT) and maximum change from baseline in ALT in all subjects | days -1, 13, 14, 16, 18, 20, 22, 24, 26, 28, follow up
Clinical safety data from spontaneous adverse event reporting, 12-lead ECG recording, vital sign measurement, nursing/physician observation and safety laboratory examination. | days -1, 13, 14, 16, 22, 26, 28, follow up
Analysis of LPS induction of IL-1b, IL-6, IL-8 and TNFa, as well as additional biomarkers, as data permit. | day 1, 14, 21, 28

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Dallas, Texas, United States